CLINICAL TRIAL: NCT06768918
Title: Digitizing Cancer Rehabilitation During and After Systemic Treatment: Feasibility Testing Implementation in South Baltic Countries
Acronym: AMBeR eRehab
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zealand University Hospital (Other)
Collaborators: Klaipėda University (Other); University of Rostock (Other); Angelholm Hospital (Other); University Clinical Centre, Gdansk (Other)
Responsible Party: Principal Investigator, Susanne Dalton, Professor, Zealand University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: p-2024-17503
Record Dates: First submitted 2024-11-27; First posted 2025-01-10 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Cancer Rehabilitation; Cancer
Keywords: Remote physical rehabilitation; cancer rehabilitation; e-health; implementation; feasibility; acceptability; exercise; physiotherapy; home-based; oncology; usability
MeSH Terms: conditions — Neoplasms; Motor Activity | interventions — Physical Therapy Modalities; Exercise; Rehabilitation

STUDY DESIGN:
Intervention Model Description: This study is a multinational multisite feasibility study of the implementation of digitally supported physical rehabilitation in five South Baltic countries (DK, PL, GER, SWE, LTU) during systemic treatment (feasibility study 1) and after systemic treatment (feasibility study 2). The feasibility studies will be run as one-arm intervention studies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Digital physical rehabilitation (Experimental): Feasibility testing the implementation of digitally delivered physical rehabilitation a) during systemic anticancer treatment and b) after completion of systemic anticancer treatment
  Interventions: Other: remote physical rehabilitation

INTERVENTIONS:
Other: remote physical rehabilitation — In this multisite international study, we feasibility test implementation of 4 different digital solutions for delivering interactive physical rehabilitation during or after systemic anticancer treatment. The contents of the intervention follows international recommendations for exercise during or after treatment for cancer.
  Other Names: physiotherapy; exercise; rehabilitation; e-rehabilitation

SUMMARY:
Background

With increasing cancer incidence and advanced cancer treatment, the growing population of cancer survivors increases the demand on health resources worldwide. Over the last 20 years, physical rehabilitation has reached recognition as an essential component of cancer care due its effect on physical function, side effects of treatment, and quality of life. However, highly specialized health care can result in longer distances to rehabilitation facilities. Also, a heavy appointment schedule for patients in treatment tends to complicate participation in rehabilitation. Telehealth has shown promise in increasing accessibility to services, also rehabilitation. However, barriers to participating in digitally delivered rehabilitation might exist, including lower e-health literacy and internet access in rural areas. The aim of this study is therefore, to examine the feasibility of implementing digitally supported rehabilitaiton in cancer care during and after treatment.

Methodology In a multinational implementation study, the feasibility of implementation of digital rehabilitation will be tested in five South Baltic Countries (DK, SWE, GER, PL, LTU). Each site will host one feasibility trial for patients during cancer treatment and one for patients after, with n=30 patients in each fesibility trial (total n=300). The intervention will be needs-based, follow international guidelines, last from 8-16 weeks, and be delivered by trained Health Care Professionals (HCP's), either fully or partially digital. Mixed methods will be used to assess outcomes of reach, effectiveness, adoption, implementation and maintenance (RE-AIM).

Through the coordinated feasibility trials across five South Baltic countries, the investigators expect to learn about important factors in implementation of digitally delivered rehabilitation in different settings, cultures, and health systems. Finally, the investigators will bring recommendations for improving reach, implementation, and sustainability of digitally delivered rehabilitation across different settings.

DETAILED DESCRIPTION:
Detailed Description

Introduction

Increasing survival rates in cancer patients has put an increasing focus on physical rehabilitation in survivorship. Physical rehabilitation plays an important role in the cancer care continuum by improving Quality of Life, functional ability and participation in everyday life. Often, however, patients may be unable to participate due to barriers related to resources, social support, distance to facility, a heavy treatment schedule and dealing with side- or late effects of treatment. Physical rehabilitation during primary, neoadjuvant or adjuvant oncological treatment could prevent loss of muscle strength, maintain or even improve physical fitness, alleviate acute toxicities of chemotherapy like fatigue, pain, depression and nausea. When entering the survivorship phase, it is also well-documented that survivors have difficulties meeting recommendations for physical activity, and the negative consequences are reduced survival and increase risk of lifestyle diseases and systemic late effects after treatment. Although physical rehabilitation is already recommended in international clinical guidelines, it is far from implemented broadly. Further, current studies indicate that there is socioeconomic inequality in who participates in the rehabilitation on offer. One reason might be the rurality of certain regions, costing patients many resources in i.e. transportation. Other reasons may include lack of resources to participate, both timewise, but also related to psychological, physical and social demands. Digital solutions may be beneficial in solving many of the barriers to participation and be a way to deliver "precision rehabilitation"; the right mode and dose to individual patients, taking personal preference and resources into consideration and utilizing them.

This study aims to feasibility test implementation of digital rehabilitation in 5 rural countries in the South Baltic.

Methods

Trial design This study is a multinational multisite feasibility study of the implementation of digitally supported physical rehabilitation in five South Baltic countries (DK, PL, GER, SWE, LTU) during systemic treatment (feasibility study 1) and after systemic treatment (feasibility study 2). The feasibility studies will be run as one-arm intervention studies.

Study setting and organization The current study is part of the Interreg South Baltic Program-funded project "AMBeR" (Advanced Modelling of Baltic cancer e-caRe). A total of seven partners from five countries are involved and are working on five different WP's. The following 5 of the 7 project partners are involved in the study (WP 4) are described here: 1) Angelholm Hospital, Region Scania, Sweden; 2) University Medical Center Rostock, Germany; 3) University Clinical Center Gdansk, Poland; 4) Klaipeda University, Lithuania; and 5) Zealand University Hospital, Denmark.

Each site will participate in the feasibility studies with á n=30:

1. early rehab (during systemic cancer treatment)
2. rehab@home (after completion of systemic cancer treatment).

Inclusion criteria

* ≥ 18 years
* Diagnosed with cancer (IDC: C00* - C97*)

Additionally, in feasibility study 1 (early rehab):

Participants should receive any systemic chemo/immunotherapy preferably (but not necessarily) with a duration of 8 weeks or more. Recruitment should be at earliest convenience preferably (but not necessarily) within 4 weeks of treatment initiation.

In feasibility study 2 (rehab@home):

Participants should preferably have completed chemotherapy/immunotherapy no more than 6 months ago but may be receiving long-standing maintenance and life-prolonging chemo-/immunotherapy.

Eligible patients are patients that have physical or psychological rehabilitation needs and that would normally be referred to physiotherapy or similar exercise specialist in cancer care, either as per normal practice or according to international guidelines.

Eligible health Care professionals delivering the intervention are those who according to local practice and authorization deliver usual care to the target groups specific to each site.

Choosing a digital solution Health care professionals/physiotherapists and the local study group at each site will be involved in choosing the digital solution to be implemented, and each site will select a unique digital solution to meet their criteria and needs. The selection is based on availability on the local market, targeted population, language availability, objectivity of movement feedback, possibility for interaction, and features for progression and regression of treatment programme. Further the demands for integrating the solution into existing IT systems is also considered. The advantages/disadvantages and costs will be weighed before a solution is selected.

Implementation

* describing the existing care process and identifying stakeholders.
* describing new care process, stakeholders and pathways in the new practice.
* Workshop 1:" setting the scene" context mapping, barriers and facilitators, solution design, action plan. Participation from all relevant stakeholders identified through context mapping of the care process. A patient representative will be involved and engaged in workshop if at all possible, and thereby contribute with the patient perspective on barriers and facilitators.
* Education and preparing HCP's in use of the digital technology and integrating it into the "toolbox" and a new professional identity.
* Workshop 2 "facilitating/supporting the ongoing process" mid-study, dealing with challenges, adjusting design, plan and support further implementation.
* Workshop 3 "picking the fruits of best practice" post-study, including examining learnings from the feasibility studies and evaluating finalized, ongoing and planed implementation.
* A logbook describing the process, actions and rationale of all steps of the implementation will be used for documentation throughout the intervention phase.

Following workshop 1, pre-study identification of expected barriers and facilitators for patients to engage in remote physical rehabilitation will be carried out through 4 steps:

1. Summary from literature review and past experience.
2. Matching most important barriers with strategies using the ERIC matching tool
3. Ranking strategies according to effectiveness and importance in the clinical setting each site by members of the study team across sites
4. Building on strategies to make action plans for implementation of the intervention each site.

Assessing Patient's and HCP's perspectives on determinants

Towards the final phase of completing the feasibility studies, the perspectives of patients' and HCP's on the important determinants for engagement in remote physical rehabilitation will be examined, applying the technique of Group Concept Mapping. The process will follow 5 pre-described steps and all activity will be online utilizing the software "GroupwisdomTM":

1. Brainstorming
2. and 3) Sorting, labelling and rating

4) Generating a cluster rating map 5) Validation of the cluster rating map The process will be performed separately for patients and HCPs, inviting a representative sample of patients for one study and all participating Intervention delivering HCP´s for a second study. For the study where patients participate, there will be a translation process of all texts and prompts to the patients' own language and back again, for the researchers to process and analyze.

Quantitative outcomes The RE-AIM framework will be used for a systematic quantification of outcomes. A range of different outcomes, measurement methods and data sources will be used as outlined in outcome measures section. For the questionnaire all partners will translate a common questionnaire into their own language using a forward-backward translation process and pilot-testing the translated questionnaire on 5-8 patients.

Data collection and management A REDCap database will be created for all study outcomes and relevant data to be collected and safely stored.

All HCP's involved in data collection will undergo a thorough training and standardization program involving physical testing, patient-reported outcome collection, recording /database familiarization, and update on international clinical guidelines in cancer rehabilitation. Monthly audits will be carried out to secure rigorous data collection is homogeneous and follows protocol.

Participant and Non-participant questionnaires To obtain information about eligible patients who decline participation in remote physical rehabilitation, decliners will be invited to answer a short questionnaire, reporting on their characteristics, reasons for refusal and barriers for participation (see table 1, decliners). Those who accept participation will receive a larger questionnaire reporting further on Patient Reported Outcome Measures (PROMs) and Acceptability. PROMs and Acceptability scales outlined in Table 1 will be collected using validated questionnaires. If not available in the local language, a forward-backward translation will be carried out and validated in 2-4 patients.

Effectiveness evaluation At the initial consultation with a HCP, the patient and HCP together will set realistic goals for the intervention, using the Patient Specific Functional Scale (PSFS) to quantify meaningful functional goals relevant to the individual patient. As per usual care, these goals may be adjusted along the way according to the patient's health status development, and the number of times adjusted will be recorded in the database. At the beginning and the end of the intervention, the patient rates themselves on a 0-10 scale how close to reaching the goal they are, and a within-patient change score will be calculated.

Harms and drop-outs An ongoing and systematic registration of harms, drop-outs and reasons for drop-out, as well as if any of the aforementioned events are likely to be associated to the delivery method of the intervention will be recorded in the database on a day-to-day basis.

Economic/resource evaluation An economic analysis will be performed using collected process data evaluating time and resources used for the remote digital rehabilitation. Data in this evaluation will cover Administrative time and contact attempts, consultation time, physiotherapist/HCP's time used in preparation/tracking the patient progress, and patients transport time (saved).

Sample size in the feasibility trials Sample size of the feasibility trials was estimated based on considerations on ensuring sufficient gathering of experiences each site, backed up by literature on recommendations for sample size in pilot trials and feasibility studies. The decision from the consortium was 30 participants each site for each feasibility study, giving a total pooled sample of 30 participants x 2 feasibility studies x 5 sites = 300 participating patients in total. The number needed to screen and invite at each site will therefore be varying and these numbers will be recorded.

Relevant concomitant care Participants will be allowed to attend concomitant usual care supplemental rehabilitation for diagnosis specific needs that cannot be met by the involved health professional or with the digital tool selected. If a participant wishes to receive usual care instead of the intervention with digital rehabilitation, they will be put on the waiting list for that.

Statistical methods Mainly descriptive statistics will be used to analyze quantitative outcomes, although effectiveness will be assessed with a pre-post change score.

Ethics approval and consent to participate Ethics approval will be applied for in each participating country with local adaptions of this protocol.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with cancer (IDC: C00* - C97*)
* Feasibility study 1 (early rehab): Participants should receive any systemic chemo/immunotherapy preferably (but not necessarily) with a duration of 8 weeks or more. Recruitment should be at earliest convenience preferably (but not necessarily) within 4 weeks of treatment initiation.
* Feasibility study 2 (rehab@home): Participants should preferably have completed chemotherapy/immunotherapy no more than 6 months ago but may be receiving long-standing maintenance and life-prolonging chemo-/immunotherapy.

Exclusion Criteria:

- Cognitively unable to give consent to, or participate in, a digital rehabilitation programme as judged by project team staff.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-03-19 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Patient's and therapist perspectives on determinants | Patients: between 4 and 12 weeks of intervention participation. Therapists: between 5 patient treatments completed and end of study (on average 1 year).
  2 Qualitative analyses using online Group Concept Mapping will be performed. One with 5-10 patients in their final phase of the rehabilitation program (minimum 1 participant each country), and one with 5-10 therapists/health professionals (minimum one each country). One -two promps phrased to create responses from informants about what the determinants are for engaging in digital e-rehabilitation, will be specified by the project group in collaboration. The process will further follow 5 pre-described steps of online activities, utilizing the software "GroupwisdomTM", The steps are as follows: Step 1) Brainstorming the prompt(s) Steps 2 and 3) Sorting, labelling and rating Step 4) Generating a cluster rating map Step 5) Validation of the cluster rating map We will perform the process separately for patients and therapists.

OTHER OUTCOMES:
Educational level | Baseline
  International Standard Classification of Education (ISCED) ISCED 0 = Early childhood education ISCED 1 = Primary Education ISCED 2 = Lower Secondary Education ISCED 3 = Upper Secondary Education ISCED 4 = Post-secondary non-Tertiary Education ISCED 5 = Short-cycle tertiary education ISCED 6 = Bachelors degree or equivalent tertiary education level ISCED 7 = Masters degree or equivalent tertiary education level ISCED 8 = Doctoral degree or equivalent tertiary education level
Employment status | baseline
  a) Full time, b) part time, c) self-employed, d) unemployed seeking work, e) unemployed not seeking work, f) student, g) retired, h) unable to work, i) other.
Attendance rates | baseline to end intervention (8-12 weeks)
  Number of attended/performed sessions versus number of prescribed sessions
Recruitment and referral rates | Baseline
  Number of referrals, number of enrolled vs. declined.
Adherence | Baseline to end of intervention (8-12 weeks)
  Exercise volume in realtion to exercise prescription
Number of monthly physical encounters between patient and therapist | During intervention (8-12 weeks)
  Fidelity to protocol: should not exceed to physical encounters per month
Health technology readiness | Assessed at one timepoint at inclusion into the study, before initiation of the intervention.
  The Readiness and enablement index for Health technology (READHY) before initiation of the intervention. (In the countries where a validated translation does not exist, one of the following will be used instead: The health education impact questionnaire (Hei-Q), The Health litteracy questionnaire (HLQ) or the eHealth Literacy Questionnaire (eHLQ), which are the scales from which the READHY items are drawn)
Barriers for participation | Baseline
  Qualitative assessment of reasons for refusal, and rural/remote-specific barriers enrolled/decliners.
Safety | During intervention (8-12 weeks)
  Registration of adverse events throughout the intervention
Acceptability | Post intervention
  Assessed by the Theoretical Framework of Acceptability (TFA)
Time consumption per patient | During intervention (8-12 weeks).
  Minutes spent in patient management, either during consultation, online or in-person, and in contact attempts.
Patient Specific Function Scale | Assessed pre- and post-intervention
  Patients own rehabilitation goal
European Organization of Research and Treatment in Cancer, core module (C30) | Assessed pre- and post-intervention (8-12 weeks)
  Health Related Quality of Life
European Organization of Research and Treatment in Cancer, fatigue module (FA12) | Assessed pre- and post-intervention (8-12 weeks)
  Validated scale for assessing fatigue in patients with cancer
EQ-5D-5L | Assessed pre- and post-intervention (8-12 weeks)
  EQ-5D_5L is a standardised measure of health-related quality of life developed by the EuroQol Group to provide a simple, generic questionnaire.
Step count, daily average | Assessed pre- and post-intervention (8-12 weeks)
  Physical activity. For the participating countries, where the digital solution for rehabilitation delivery does not measure step counts, the Godin Shephard Leisure Time Questionnaire or the International Physical Activity Questionnaire will be used to assess physical activity instead.
Gait speed | Assessed pre- and post-intervention (8-12 weeks)
  4- or 10-meters speed test, accoding to local availability/space
30 second sit-to-stand | Assessed pre- and post-intervention (8-12 weeks)
  Physical function; number of sit to stand repetitions in 30 seconds.
Timed up and go | Assessed pre- and post-intervention (8-12 weeks)
  Physical function alternative test
Hand grip strength | Assessed pre- and post-intervention (8-12 weeks)
  Hand grip dynamometry: in Newton.
Tandem test | Assessed pre- and post-intervention (8-12 weeks)
  Balance
6-minute walk test | Assessed pre- and post-intervention (8-12 weeks)
  Endurance
Watt max test | Assessed pre- and post-intervention (8-12 weeks)
  Endurance alternative test
Cancer disease | baseline
  Cancer type, cancer treatment, treatment intent.
Body height | baseline
  measured in meters
Body weight | baseline
  Measured in kilograms

CONTACTS AND LOCATIONS:
Overall Officials: Susanne O Dalton, MD PhD, Principal Investigator — Zealand University Hospital, Department of Clinical Oncology and Palliative Care
Locations (5):
- Zealand Unievrsity Hospital, Næstved, Denmark
- University Medical Center Rostock, Rostock, Germany
- Klaipeda University, Klaipėda, Lithuania
- Medical University of Gdansk, Gdansk, Poland
- Ängelholm Hospital, Ängelholm, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
This study classifies in the domain of implementation studies, and therefore the focus of interest is on implementation data and not on individual particpant data. Whether the data will be suitable for sharing has not yet been discussed and depends on national regulations in each participating country.

REFERENCES:
- [Background] Totton N, Lin J, Julious S, Chowdhury M, Brand A. A review of sample sizes for UK pilot and feasibility studies on the ISRCTN registry from 2013 to 2020. Pilot Feasibility Stud. 2023 Nov 21;9(1):188. doi: 10.1186/s40814-023-01416-w. PMID 37990337
- [Background] Stratford P, Gill C, Westaway M, Binkley J. Assessing disability and change on individual patients: a report of a patient specific measure. Physiotherapy Canada. 1995(47):258-63.
- [Background] Glasgow RE, Vogt TM, Boles SM. Evaluating the public health impact of health promotion interventions: the RE-AIM framework. Am J Public Health. 1999 Sep;89(9):1322-7. doi: 10.2105/ajph.89.9.1322. PMID 10474547
- [Background] Trochim WM, McLinden D. Introduction to a special issue on concept mapping. Eval Program Plann. 2017 Feb;60:166-175. doi: 10.1016/j.evalprogplan.2016.10.006. Epub 2016 Oct 11. PMID 27780609
- [Background] Powell BJ, Waltz TJ, Chinman MJ, Damschroder LJ, Smith JL, Matthieu MM, Proctor EK, Kirchner JE. A refined compilation of implementation strategies: results from the Expert Recommendations for Implementing Change (ERIC) project. Implement Sci. 2015 Feb 12;10:21. doi: 10.1186/s13012-015-0209-1. PMID 25889199
- [Background] Ryan M, Lam N, Wright K, Siderov J. Clinical Oncology Society of Australia Position Statement: 2022 update to the safe handling of monoclonal antibodies in healthcare settings. Asia Pac J Clin Oncol. 2023 Dec;19(6):723-730. doi: 10.1111/ajco.13943. Epub 2023 Mar 10. PMID 36899469
- [Background] Sweegers MG, Altenburg TM, Chinapaw MJ, Kalter J, Verdonck-de Leeuw IM, Courneya KS, Newton RU, Aaronson NK, Jacobsen PB, Brug J, Buffart LM. Which exercise prescriptions improve quality of life and physical function in patients with cancer during and following treatment? A systematic review and meta-analysis of randomised controlled trials. Br J Sports Med. 2018 Apr;52(8):505-513. doi: 10.1136/bjsports-2017-097891. Epub 2017 Sep 27. PMID 28954800
- [Background] Ibeggazene S, Turner R, Rosario D, Bourke L. Remote interventions to improve exercise behaviour in sedentary people living with and beyond cancer: a systematic review and meta-analysis. BMC Cancer. 2021 Mar 24;21(1):308. doi: 10.1186/s12885-021-07989-0. PMID 33761906
- [Background] Felser S, Behrens M, Lampe H, Henze L, Grosse-Thie C, Murua Escobar H, Rohde K, Albrecht I, Zschorlich V, Junghanss C. Motivation and preferences of cancer patients to perform physical training. Eur J Cancer Care (Engl). 2020 Jul;29(4):e13246. doi: 10.1111/ecc.13246. Epub 2020 May 31. PMID 32476203
- [Background] Davies JM, Sleeman KE, Leniz J, Wilson R, Higginson IJ, Verne J, Maddocks M, Murtagh FEM. Socioeconomic position and use of healthcare in the last year of life: A systematic review and meta-analysis. PLoS Med. 2019 Apr 23;16(4):e1002782. doi: 10.1371/journal.pmed.1002782. eCollection 2019 Apr. PMID 31013279
- [Background] Kennedy MA, Bayes S, Newton RU, Zissiadis Y, Spry NA, Taaffe DR, Hart NH, Galvao DA. Implementation barriers to integrating exercise as medicine in oncology: an ecological scoping review. J Cancer Surviv. 2022 Aug;16(4):865-881. doi: 10.1007/s11764-021-01080-0. Epub 2021 Sep 12. PMID 34510366
- [Background] Cormie P, Atkinson M, Bucci L, Cust A, Eakin E, Hayes S, McCarthy S, Murnane A, Patchell S, Adams D. Clinical Oncology Society of Australia position statement on exercise in cancer care. Med J Aust. 2018 Aug 20;209(4):184-187. doi: 10.5694/mja18.00199. Epub 2018 May 7. PMID 29719196
- [Background] Ligibel JA, Bohlke K, May AM, Clinton SK, Demark-Wahnefried W, Gilchrist SC, Irwin ML, Late M, Mansfield S, Marshall TF, Meyerhardt JA, Thomson CA, Wood WA, Alfano CM. Exercise, Diet, and Weight Management During Cancer Treatment: ASCO Guideline. J Clin Oncol. 2022 Aug 1;40(22):2491-2507. doi: 10.1200/JCO.22.00687. Epub 2022 May 16. PMID 35576506
- [Background] Patel AV, Friedenreich CM, Moore SC, Hayes SC, Silver JK, Campbell KL, Winters-Stone K, Gerber LH, George SM, Fulton JE, Denlinger C, Morris GS, Hue T, Schmitz KH, Matthews CE. American College of Sports Medicine Roundtable Report on Physical Activity, Sedentary Behavior, and Cancer Prevention and Control. Med Sci Sports Exerc. 2019 Nov;51(11):2391-2402. doi: 10.1249/MSS.0000000000002117. PMID 31626056
- [Background] Lahart IM, Metsios GS, Nevill AM, Carmichael AR. Physical activity, risk of death and recurrence in breast cancer survivors: A systematic review and meta-analysis of epidemiological studies. Acta Oncol. 2015 May;54(5):635-54. doi: 10.3109/0284186X.2014.998275. Epub 2015 Mar 9. PMID 25752971
- [Background] Campbell KL, Winters-Stone KM, Wiskemann J, May AM, Schwartz AL, Courneya KS, Zucker DS, Matthews CE, Ligibel JA, Gerber LH, Morris GS, Patel AV, Hue TF, Perna FM, Schmitz KH. Exercise Guidelines for Cancer Survivors: Consensus Statement from International Multidisciplinary Roundtable. Med Sci Sports Exerc. 2019 Nov;51(11):2375-2390. doi: 10.1249/MSS.0000000000002116. PMID 31626055
- [Background] Andersen HH, Vinther A, Lund CM, Paludan C, Jorgensen CT, Nielsen D, Juhl CB. Effectiveness of different types, delivery modes and extensiveness of exercise in patients with breast cancer receiving systemic treatment - A systematic review and meta-analysis. Crit Rev Oncol Hematol. 2022 Oct;178:103802. doi: 10.1016/j.critrevonc.2022.103802. Epub 2022 Aug 27. PMID 36031174
- See also: Homepage for the AMBeR project, of which the AMBeR eRehab is a work package and separately registered study. — https://amber.ku.lt/en/advanced-modeling-of-baltic-cancer-e-care-amber